CLINICAL TRIAL: NCT02464761
Title: Photodynamic Therapy (PDT) for the Treatment of Vertebral Metastases: A Prospective Phase I Clinical Trial
Brief Title: Photodynamic Therapy for the Treatment of Vertebral Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Albert Yee, Orthopaedic Surgeon, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT01
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Vertebral Metastases
MeSH Terms: interventions — Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalating PDT (Experimental)
  Interventions: Drug: Visudyne

INTERVENTIONS:
Drug: Visudyne
  Other Names: Verteporfin

SUMMARY:
An estimated 10 percent of primary breast, prostate, lung, thyroid and renal cell tumors metastasize to the spine. The majority of these tumors are detected before surgical intervention is required and most patients receive radiation therapy for symptomatic relief. Complete pain control, duration of pain control, high recurrence rates and soft tissue complications make radiation a less than ideal treatment. Also, pre-operative radiation therapy is a significant negative predictor for surgical outcomes. To improve the treatment options for patients with advanced cancer with spinal lesions the research team investigated a new minimally invasive therapy known as photodynamic therapy (PDT) that targets metastatic spine lesions with limited side effects. PDT involves the use of a photo-activated chemotherapeutic agent, given intravenously that when stimulated by non-thermal wavelength-specific light allows for selective ablation of tumor tissue. The light is delivered to the spine through small fiber optic cables using a diode laser. By combining canine and porcine studies the investigators have strong evidence to support that PDT is both safe and effective for the treatment of metastatic tumors in the spine. PDT is targeted, repeatable, minimally invasive and has limited local and systemic side effects. Its use would enhance the treatment options for patients with advanced stage cancer. The goal of the present study is to demonstrate that PDT can be safely and effectively given to treat spinal metastases in patients with advanced stage cancer who have multiple lesions or who have failed radiation or surgical intervention. The effectiveness of this treatment will be determined through clinical and radiographic endpoints along with recurrence and survival. The investigators intend to demonstrate that PDT is a minimally invasive method with low morbidity and mortality by which spinal tumors can be ablated and later stabilized through vertebroplasty, optimizing quality of life and providing effective treatment.

DETAILED DESCRIPTION:
There are over 1.5 million cases of cancer reported each year in North America and a significant number of patients eventually suffer from metastases to the spine which present as an extremely challenging problem for both the clinician and patient. Primary tumors that most commonly affect the spine include breast, prostate, lung, thyroid and renal cell cancer. Estimates from large clinical series report at least a 10 percent rate of metastases to the spine from these most common tumors. These lesions are extremely painful and significantly affect the quality of life of advanced stage cancer patients. The majority of these tumors are detected before surgical intervention is required and most patients receive radiation therapy for their spine lesions for symptomatic relief. However, complete pain control, duration of pain control along with a high recurrence rate of lesions and soft tissue complications makes radiation a less than an ideal treatment. In addition, pre-operative radiation therapy is a significant negative prognosticator for surgical outcomes.

To improve the treatment options for patients with advanced cancer with spinal lesions the research team has investigated a new minimally invasive therapy, known as photodynamic therapy (PDT) that targets metastatic spine lesions directly and has limited side effects. PDT involves the use of a photo-activated chemotherapeutic agent, benzoporphyrin derivative (verteporfin/Visudyne) given intravenously that when stimulated by non-thermal wavelength-specific light allows for selective ablation of tumor tissue. The light is delivered to the spine through small fiber optic cables (outer diameter 0.98mm, inner core of 0.5mm mm) using a diode laser. Visudyne is an FDA and Health Canada approved photosensitizer that has been used in over one million patients for the treatment of age related macular degeneration, a leading cause of blindness in the elderly. To investigate the use of PDT for spinal metastases the investigators initially developed a bioluminescent metastatic rodent model using human breast cancer that metastasized to the spine. Using this model it was determined that PDT was effective at treating metastatic breast cancer lesions in the spine. The research team next utilized non-tumor bearing canine and porcine models to determine that the treatment could be safely delivered to the spine and conduct light dosimetry analysis. The safety of PDT intra-operatively was assessed using somatosensory evoked potentials and through post-treatment clinical examination and magnetic resonance imaging (MRI). The effects PDT had on the spine were analyzed by comparing pre-operative and post-operative MR imaging and correlating those in turn with histological analysis. None of these animals suffered weakness or complication from the use of PDT around the spinal cord. During these studies the investigators developed the planning, delivery and instrumentation methodologies to deliver PDT to spinal tumors and the methodology to combine this therapy with vertebroplasty, a percutaneous method of stabilizing the spine. In addition, in a separate set of studies, highgrade osteosarcomas in canines were treated to determine the effect PDT had on large bone tumors. The results of this study again provided comparison of pre and post-treatment effects seen on MRI and histological analysis. The volume of effect seen in the osteosarcomas was up to 25cm (cubed) and was comparable to the volume of effect required for complete treatment of spinal lesions. By combining the canine and porcine studies there is strong evidence that PDT is both safe and effective for the treatment of metastatic tumors in the spine.

PDT has many advantages over current therapies; it is targeted, repeatable, minimally invasive and has limited local and systemic side effects. Its use would enhance the treatment options for patients with advanced stage cancer. The goal of the present study is to demonstrate that PDT can be safely and effectively given to treat spinal metastases in patients with advanced stage cancer. The study is a pilot study and will determine the safe and accurate treatment of 30 patients with spinal metastases who have multiple lesions or who have failed radiation or surgical intervention. The effectiveness of this treatment will be determined through clinical and radiographic endpoints with recurrence and survival also determined. The investigators intend to demonstrate that PDT provides a minimally invasive method with low morbidity and mortality by which spinal tumors can be ablated and later stabilized through vertebroplasty, optimizing quality of life and providing effective treatment for this devastating manifestation of advanced stage cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 85
* Established metastatic vertebral bony disease in the spine
* Eligible for single level vertebral osteoplasty (i.e. percutaneous vertebroplasty, kyphoplasty)
* Patients who are symptomatic with axial pain from vertebral metastatic involvement and are at risk for pathologic fracture; or have had a symptomatic pathologic fracture
* Patients who have shown radiographic progression and/or pain symptoms of a documented vertebral metastasis despite non-surgical therapies

Exclusion Criteria:

* Progressive neurological compromise
* Osteoblastic vertebral metastatic disease
* Posterior vertebral cortical/body wall involvement
* Spinal canal compromise / neurologic compression
* Anticipated life expectancy of less than twelve weeks to live
* Cognitive impairment and/or language barriers to study participation
* Severe hepatic impairment (Child's C) with active hepatitis or hepatic disease.
* Active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, requirement for corticosteroids and/or progressive growth. CNS metastases must be stable for > 2 weeks prior to screening.)
* Nursing mothers, pregnant, currently breastfeeding or trying to get pregnant.
* Unable to avoid sun exposure for 5 day post-PDT therapy (per verteporfin precautions).
* Hyperphotosensitivity conditions, including porphyria
* Hypersensitivity to verteporfin or any other ingredients of Visudyne

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative dosimetry | During surgery
  Intraoperative dosimetry data on light transmission and attenuation in patient specific diseased bone will be contrasted to pre-operative imaging data and the region of effect based on actual light transmission compared to pre-operative planning algorithms. These results will gauge the potential accuracy of our planning algorithms.

SECONDARY OUTCOMES:
Neurologic function | 7 days, 6 weeks
  The primary safety parameter will be unexpected worsening in neurological function.
  Physical examination will include a detailed neurological examination (including ASIA score) that assesses the strength, sensation and reflexes of the patient in the upper and lower extremities

OTHER OUTCOMES:
Effect of PDT and vertebral osteoplasty on patient functional outcome - SF36 | 7 days, 6 weeks
  The analgesic effect of surgical treatment will be estimated using the SF-36
Effect of PDT and vertebral osteoplasty on patient functional outcome - VAS scale | 7 days, 6 weeks
  The analgesic effect of surgical treatment will be estimated using the visual analogue (VAS) pain scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No